CLINICAL TRIAL: NCT05757999
Title: Effect of Magnesium Sulphate Pretreatment on Cis-Atracurium Induced Neuromuscular Block and Recovery Characteristics: A Randomized Controlled Trial.
Brief Title: Effect of MgSO4 Pretreatment on Muscle Relaxation
Acronym: MgSO4/CisA
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04-2023-200100
Record Dates: First submitted 2023-02-19; First posted 2023-03-07 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Muscle Relaxation
MeSH Terms: interventions — Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients will be allocated to one of two groups: a saline placebo group (n=50) or a magnesium group (n=50). The patients will be pretreated with either an intravenous 0.9% saline infusion (total volume 100 ml, infusion rate 10 ml min-1) or a magnesium sulphate infusion (60 mg kg-1, total volume 100 ml, infusion rate 10 ml min-1) 10 min. before induction of anesthesia. Allocation numbers will be placed in opaque envelopes and opened by an anesthesiologist (not participating in the study)who will also prepare the study solutions.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Allocation numbers will be placed in opaque envelopes and opened by an anesthesiologist (not participating in the study)who will also prepare the study solutions. The solutions used in the study are similar in physical appearance and an investigator not included in the study will prepare the solutions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MgSo4 (Active Comparator): A magnesium sulphate infusion (60 mg kg-1, total volume 100 ml, infusion rate 10 ml min-1) 10 min. will be administered before induction of anesthesia
  Interventions: Drug: Magnesium Sulphate
- Saline Placebo (Placebo Comparator): an intravenous 0.9% saline infusion (total volume 100 ml, infusion rate 10 ml min-1) 10 min. will be administered before induction of anesthesia.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Magnesium Sulphate — A magnesium sulphate infusion (60 mg kg-1, total volume 100 ml, infusion rate 10 ml min-1) will be administered to patients 10 min. before induction of anesthesia.
  Other Names: MgSo4
  Arms: MgSo4
Drug: Saline — The patients will be pretreated with an intravenous 0.9% saline infusion (total volume 100 ml, infusion rate 10 ml min-1) 10 min before induction of anesthesia.
  Other Names: Placebo Comparator
  Arms: Saline Placebo

SUMMARY:
In this study, the effect of magnesium sulphate on the onset and duration of intense and moderate cis-atracurium induced neuromuscular blocking and on the period of no response to nerve stimulation will be evaluated in patients who will recieve magnesium sulphate (intervention group) and patients who will not recieve magnesium sulphate (comparator group).

DETAILED DESCRIPTION:
General anesthesia is a drug-induced reversible state consisting of unconsciousness, amnesia, anti-nociception, and immobility, with maintenance of physiological stability. Balanced general anesthesia, the most common management strategy used in anesthesia care, entails administering a combination of different agents to create the anesthetic state. There is evidence that balanced general anesthesia uses less of each drug than if the drug were administered alone. This approach is believed to increase the likelihood of a drug's desired effects and reduce the likelihood of its side effects. With addition of adjuvants, Alpha-2 adrenoceptor agonists, such as dexmedetomidine, are known to possess amnesic, analgesic, sympatholytic, and antinociceptive properties, and therefore, can reduce the requirement of anesthetics and opioids intraoperatively. Administration of MgSO4 has also shown significant reduction in the perioperative requirement of propofol, opioids, and muscle relaxants. Magnesium sulphate has gained prominence as an adjuvant drug in multimodal anesthesia and pain medicine. It has several clinical indications including attenuation of the adrenergic response to tracheal intubation and improved peri-operative analgesia. Magnesium sulphate also enhances the action of non-depolarizing neuromuscular blocking drugs, resulting in potentiation of neuromuscular blockade (NMB).The site of magnesium potentiation of neuromuscular blocking drugs is the motor end plate, where magnesium reduces the release of prejunctional acetylcholine, thereby decreasing the muscle membrane excitability. However, limited data exist concerning the effect of magnesium sulphate on the duration of deep or intense NMB and on the period of no response to nerve stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Age group 18-60 years old
* Both genders
* Patients who will be scheduled to undergo elective otorhinolaryngological surgery.
* Patients with BMI between 18.5 and 24.9 Kg/m2.
* Patients with American Society of Anesthesiologist physical status classification of 1 or 2

Exclusion Criteria:

* Patients who are less than 18 years old or more than 60 years old.
* Patients on medications that interfered with muscle activity.
* Allergy to medications used in this study.
* Pregnancy or suspected pregnancy.
* Neuro-muscular diseases.
* Renal or hepatic impairment.
* Hypermagnesemia (>2.5 mmol) or hypomagnesemia (<1.7 mmol).
* Patients refusing to study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-23 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
The duration of the period of no response. | Intraoperative.
  The effect of pretreatment with magnesium sulphate on the duration of the period of no response will be measured with the TOF-Watch SX (Organon Ireland Ltd, Dublin, Ireland). The ulnar nerve near the wrist will be stimulated and the activity of the adductor pollicis (thumb) muscle will be recorded.

SECONDARY OUTCOMES:
The duration of intense neuromuscular block (minutes) | Intraoperative
  The effect of pretreatment with magnesium sulphate on the duration of the intense neuromuscular block in minutes will be measured with the TOF-Watch SX (Organon Ireland Ltd, Dublin, Ireland). The ulnar nerve near the wrist will be stimulated and the activity of the adductor pollicis (thumb) muscle will be recorded.
The duration of deep neuromuscular block | Intraoperative.
  The effect of pretreatment with magnesium sulphate on the duration of the deep neuromuscular block in minutes will be measured with the TOF-Watch SX (Organon Ireland Ltd, Dublin, Ireland). The ulnar nerve near the wrist will be stimulated and the activity of the adductor pollicis (thumb) muscle will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Hala Abdel-Ghaffar, MD, Principal Investigator — Professor of anesthesia and intensive care, faculty of medicine, Assiut university, Assiut, Egypt.
Locations (1):
- Assiut university main hospital, ENT operative theatre, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No